CLINICAL TRIAL: NCT02790320
Title: Eribulin [Halaven] Use For the Treatment of Advanced Breast Cancer: Observational Retrospective Analysis
Brief Title: Eribulin [Halaven] Use For the Treatment of Advanced Breast Cancer
Acronym: EUFORIA-1
Status: Completed | Type: Observational
Sponsor: Eisai Farmacêutica S.A. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: OBU-SW-H-01
Record Dates: First submitted 2016-05-31; First posted 2016-06-03 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-04

CONDITIONS: Metastatic Breast Cancer
Keywords: Eribulin mesylate; Halaven; Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with locally recurrent or metastatic breast cancer: Patients received 1.4 mg/m2 eribulin, administered intravenously on day 1 and 8 of each 21 day cycle until disease progression or unmanageable toxicity, per routine clinical practice.

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of eribulin in standard clinical practice in patients with locally recurrent or metastatic advanced breast cancer.

DETAILED DESCRIPTION:
This was an observational, cross-sectional, retrospective, multicenter study conducted in Spain. During the year after authorization of the drug by the European Medicines Agency (EMA), patients in the compassionate use program (public sites) and patients treated in private sites (no purchase restrictions) who received at least 1 dose of treatment with eribulin per approved label at any of the 17 Spanish sites with the highest numbers of treated cases during that period (minimum 3 patients/site) were enrolled in this observational study. Approximately 112 patients will be enrolled in the study.

ELIGIBILITY:
Inclusion criteria:

1. Patients diagnosed with locally recurrent or metastatic advanced breast cancer, previously treated with taxanes and anthracyclines, unless these were not indicated.
2. Clinical and/or radiological documentation of location and extension of the disease at the time of starting treatment with eribulin. Patients with measurable diseases and those patients who only have non-measurable lesions are eligible.
3. Medical history documentation including analytical control data (blood count and serum chemistry including hepatic and renal functions) carried out at least one week before starting treatment with eribulin. (Determining the CA15-3 tumor marker is not indispensable).
4. Eribulin monotherapy (at least 1 dose) between April 2011 and March 2012, both inclusive.
5. Availability of a medical history allowing monitoring of clinical progression of the patients during and after treatment with eribulin.

Exclusion criteria:

1. Diagnosis of any type of cancer in the last 5 years, except for non-melanoma skin cancer, cervical intraepithelial neoplasia or contralateral breast cancer.
2. Patients having received any other anti-tumor treatment, whether conventional or experimental, during the week prior to starting treatment with eribulin. Treatment with bisphosphonate and corticoids is allowed if they are clinically indicated and started 28 days before treatment with eribulin.
3. Lack of clinical status documentation after completing treatment with eribulin or, at least, after having been administered 3 initial cycles. This can arise in any of the following cases (they are not excluding):

   1. Patients whose Medical History does not state the reason and date for interruption of treatment with eribulin and their subsequent clinical progression.
   2. Patients still undergoing treatment with eribulin on March 31, 2012, for whom there is no data for at least the first 3 cycles.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally recurrent or metastatic advanced breast cancer who were treated with eribulin
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2012-06; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Clinical benefit rate | From signing of informed consent up to 1 year

SECONDARY OUTCOMES:
Objective response rate | From signing of informed consent up to 1 year
Overall survival | From signing of informed consent up to 1 year
Progression-free survival | From signing of informed consent up to 1 year
Change from baseline in tumor markers CA15-3 | Baseline and up to 1 year
Time to response from start of treatment | From signing of informed consent up to 1 year
Duration of response | From signing of informed consent up to 1 year
Duration of stabilization | From signing of informed consent up to 1 year
Post-treatment survival | From signing of informed consent up to 1 year
Progression time after interruption | From signing of informed consent up to 1 year
Number of patients with adverse events / serious adverse events | From signing of informed consent up to 1 year

CONTACTS AND LOCATIONS:
Locations (17):
- Spain (17):
  - Hospital Comarcal de Barbastro, Huesca
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital Arnau de Vilanova, Lleida
  - Clínica Román, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Madrid Norte Sanchinarro, Madrid
  - Hospital MD Anderson, Madrid
  - Hospital Quirón Madrid, Madrid
  - Hospital Sanitas La Moraleja, Madrid
  - Hospital Universitario Morales Meseguer, Murcia
  - Hospital de Navarra, Navarra
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Clínica Esperanza de Triana, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Virgen Macarena, Seville
  - Hospital Miguel Servet, Zaragoza